CLINICAL TRIAL: NCT02137278
Title: Randomized Controlled Trial on Discontinuation of Vasoactive Drugs in Patients With Hypotensive Reflex Syncope
Brief Title: Stop Vasodepressor Drugs in Reflex Syncope
Acronym: STOP-VD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano Multidisciplinare per lo Studio della Sincope (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASL4/CARD/01
Record Dates: First submitted 2014-05-01; First posted 2014-05-13 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Hypotensive Syncope
Keywords: Syncope; Presyncope; Vasoactive drugs; Hypotension; Carotid sinus massage; Tilt table test
MeSH Terms: conditions — Syncope; Hypotension | interventions — Antihypertensive Agents; Nitrates; Diuretics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stop/reduce vasoactive drugs (Active Comparator): Discontinuation of any vasoactive therapy or reduction of vasoactive drug therapies as much as possible according to clinical judgment
  Interventions: Other: Stop/reduce vasoactive drugs
- Vasoactive drug therapy (Experimental): Continue current vasoactive therapy
  Interventions: Drug: Vasoactive drug therapies

INTERVENTIONS:
Drug: Vasoactive drug therapies — Continue current vasoactive therapy
  Other Names: Antihypertensive; Nitrates; Alpha-antagonists; Diuretics; Neuroleptic antidepressant; L-dopa antagonists
  Arms: Vasoactive drug therapy
Other: Stop/reduce vasoactive drugs — Discontinuation of any vasoactive therapy or reduction of vasoactive drug therapies as much as possible according to clinical judgment.
  Other Names: Antihypertensive; Nitrates; Alpha-antagonists; Diuretics; Neuroleptic antidepressant; L-dopa antagonists
  Arms: Stop/reduce vasoactive drugs

SUMMARY:
Investigate clinical effects (reduction of number of syncope and associate symptoms) of suspension of vasoactive drugs in patients affected by vasodepressor reflex syncope.

DETAILED DESCRIPTION:
Several drugs which are commonly used in clinical practice, such as antihypertensive, antiarrhythmic and psychiatric drugs, are associated with orthostatic hypotension and syncope. This phenomenon is much more evident in the elderly and with multiple therapies. The present study was aimed to investigate, in patients affected by reflex syncope, the clinical effects (reduction in syncope recurrence and associated symptoms) and the laboratory tests (negativization of carotid sinus massage and tilt table test) when such drugs are discontinued or reduced

ELIGIBILITY:
Inclusion Criteria:

Patients assuming chronic (>1 year) vasoactive therapy affected by reflex recurrent (>2 episodes) syncopes who have a positive dominant vasodepressor or mixed response to tilt table test and/or carotid sinus massage

Exclusion Criteria:

1. Orthostatic hypotension defined as fall in systolic blood pressure >20 mmHg during the first 3 minutes of active standing
2. Competing diagnosis of syncope different from hypotensive reflex syncope
3. Reflex syncope with negative response to carotid sinus massage and tilt table test
4. Cardioinhibitory reflex syncope which requires permanent cardiac pacing
5. Severe hypertension which requires treatment (>150/95)
6. Structured heart disease which requires hypotensive therapy in order to prevent acute heart failure
7. Cardiac hypotensive therapy in order to prevent recurrences
8. Previous stroke or transient ischemic attacks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Recurrence of syncope or presyncope and adverse events | From date of randomization until the date of first documented syncope or adverse event, whichever came first, assessed up to 2 years
  Combined end-point of rate of patients with recurrence of (pre)syncope and adverse events

SECONDARY OUTCOMES:
Syncope | From date of randomization until the date of first documented syncope or adverse event, whichever come first, assessed up to 2 years
  Recurrence of syncope
Presyncope | From date of randomization until the date of first documented syncope or adverse event, whichever came first, assessed up to 2 years
  Burden of presyncope, measured as number of episodes of presyncope/s per month assessed up to 2 years by mean of a patient's diary

OTHER OUTCOMES:
Acute study | 1 month
  Quality of life assessed by means of the Specific symptom Scale - Orthostatic Hypotension questionnaire. Results of carotid sinus massage and tilt table test

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento di Cardiologia, Ospedali del Tigullio, Lavagna, Italy

REFERENCES:
- [Background] Gaggioli G, Brignole M, Menozzi C, Devoto G, Oddone D, Gianfranchi L, Gostoli E, Bottoni N, Lolli G. A positive response to head-up tilt testing predicts syncopal recurrence in carotid sinus syndrome patients with permanent pacemakers. Am J Cardiol. 1995 Oct 1;76(10):720-2. doi: 10.1016/s0002-9149(99)80207-0. No abstract available. PMID 7572635
- [Result] Solari D, Maggi R, Oddone D, Solano A, Croci F, Donateo P, Brignole M. Clinical context and outcome of carotid sinus syndrome diagnosed by means of the 'method of symptoms'. Europace. 2014 Jun;16(6):928-34. doi: 10.1093/europace/eut283. Epub 2013 Sep 20. PMID 24058183
- [Result] Podoleanu C, Maggi R, Brignole M, Croci F, Incze A, Solano A, Puggioni E, Carasca E. Lower limb and abdominal compression bandages prevent progressive orthostatic hypotension in elderly persons: a randomized single-blind controlled study. J Am Coll Cardiol. 2006 Oct 3;48(7):1425-32. doi: 10.1016/j.jacc.2006.06.052. Epub 2006 Sep 14. PMID 17010806
- [Result] Brignole M, Menozzi C, Gaggioli G, Musso G, Foglia-Manzillo G, Mascioli G, Fradella G, Bottoni N, Mureddu R. Effects of long-term vasodilator therapy in patients with carotid sinus hypersensitivity. Am Heart J. 1998 Aug;136(2):264-8. doi: 10.1053/hj.1998.v136.89911. PMID 9704688